CLINICAL TRIAL: NCT07034157
Title: A Real-World Study on Ultrasound-Based Screening and Integrated Therapeutic Strategies for Patients With Concomitant Coronary and Cervicocephalic Artery Stenosis
Acronym: ANGEL-UNIFY
Status: Recruiting | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Xiaochuan Huo, Prof, Beijing Anzhen Hospital
Other Study IDs: KS2025006
Record Dates: First submitted 2025-06-15; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Coronary Artery Disease; Carotid Artery Stenosis; Cerebrovascular Disorders
Keywords: Coronary Artery Disease; Carotid Artery Stenosis; Doppler Ultrasound; Combined Vascular Intervention
MeSH Terms: conditions — Coronary Artery Disease; Carotid Stenosis; Cerebrovascular Disorders | interventions — Percutaneous Coronary Intervention; Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: PCI + Carotid Revascularization: Patients diagnosed with both coronary artery disease and significant carotid artery stenosis requiring intervention, who received both PCI and carotid revascularization.
  Interventions: Procedure: Percutaneous Coronary Intervention; Procedure: Cerebrovascular Intervention (CAS ）
- Group 2: PCI + Observation of Carotid Stenosis: Patients who underwent PCI for coronary artery disease, with no carotid stenosis or with carotid stenosis not requiring or not receiving interventional treatment.
  Interventions: Procedure: Percutaneous Coronary Intervention; Other: No Intervention / Observation
- Group 3: Observation Only (No PCI + No CAS): Patients who did not undergo PCI and either had no carotid artery stenosis or were managed medically for carotid stenosis without any revascularization.
  Interventions: Other: No Intervention / Observation

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention — Coronary stenting performed as part of routine care for patients with coronary artery stenosis.
  Groups: Group 1: PCI + Carotid Revascularization; Group 2: PCI + Observation of Carotid Stenosis
Procedure: Cerebrovascular Intervention (CAS ） — Patients with intervention-indicated head and neck artery stenosis will receive carotid artery stenting based on clinical evaluation.
  Groups: Group 1: PCI + Carotid Revascularization
Other: No Intervention / Observation — Clinical observation or standard follow-up in patients without significant disease
  Groups: Group 2: PCI + Observation of Carotid Stenosis; Group 3: Observation Only (No PCI + No CAS)

SUMMARY:
This prospective observational cohort study aims to investigate the prevalence and clinical significance of head and neck arterial stenosis in patients with coronary artery disease (CAD) undergoing or scheduled for percutaneous coronary intervention (PCI). Using Doppler ultrasound as the primary screening tool, the study will assess the degree of stenosis and evaluate the impact of different combined treatment strategies on patient outcomes. The research will provide real-world evidence to optimize integrated care approaches for patients with comorbid cardiovascular and cerebrovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Patients with coronary artery disease scheduled to undergo elective percutaneous coronary intervention (PCI) on the following day.

Exclusion Criteria:

1. The expected survival is less than 1 years;
2. Simultaneously merge other serious diseases;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (aged ≥18 years) diagnosed with coronary artery stenosis who are scheduled for or have recently undergone percutaneous coronary intervention (PCI), and who will undergo ultrasound screening for concomitant head and neck arterial stenosis. Participants will be enrolled from a tertiary care hospital in China as part of a prospective observational cohort.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Head and Neck Artery Stenosis in Patients with Coronary Artery Disease | At baseline (prior to or during initial hospitalization)
  The proportion of patients with coronary artery disease who are found to have head and neck artery (e.g., carotid or vertebral artery) stenosis, as determined by duplex ultrasound or other imaging modalities.

SECONDARY OUTCOMES:
mRS score | 7±1 days or the day discharged
mRS Score | 90±7 days
mRS Score | 365±30 days
Rate of cardiovascular and cerebrovascular events | 90±7 days
Rate of cardiovascular and cerebrovascular events | 365±30 days
Short-term complications | 90±7 days
Long-term complications | 365±30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No